CLINICAL TRIAL: NCT03233542
Title: The Association Between Physical Sensations and Thinking Styles [Der Zusammenhang Zwischen körperlichem Empfinden Und Denkstilen]
Brief Title: The Association Between Physical Sensations and Thinking Styles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Collaborators: German Research Foundation (Other); University of Oxford (Other); University of Salzburg (Other)
Responsible Party: Principal Investigator, Marcella Woud, Postdoctoral Research Fellow, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 145; WO2018/2-1 (Other Grant/Funding Number: Deutsche Forschungsgemeinschaft (DFG)); MA1116/13-1 (Other Grant/Funding Number: Deutsche Forschungsgemeinschaft (DFG))
Record Dates: First submitted 2017-07-23; First posted 2017-07-28 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Panic Disorder
Keywords: Cognitive biases; Associations; Interpretations; Physiological and biological markers
MeSH Terms: conditions — Panic Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants meeting study criteria for Panic Disorder will be randomized to an intervention arm (CBT) or waiting list arm (which is followed by CBT after completion of the study procedures); participants meeting study criteria for the anxious control group will be allocated to an intervention (CBT) arm. The study aims to have equal numbers of participants in each of the 3 arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Panic Disorder: CBT (Experimental): Participants with Panic Disorder randomized to this arm will receive a manualised Cognitive Behaviour Therapy (CBT) treatment for Panic Disorder, delivered in the outpatient psychotherapy centre of the Department of Clinical Psychology and Psychotherapy, Ruhr-Universität Bochum.
  Interventions: Behavioral: Cognitive Behaviour Therapy
- Panic Disorder: Waiting list (No Intervention): After the pre-treatment testing session, participants with Panic Disorder randomized to this arm will wait a length of time equivalent to that for the pre/post-treatment duration for the Panic Disorder: Cognitive Behaviour Therapy arm (approx. 3 months), before returning to the post-treatment assessment. After completing all the study procedures, participants in this arm receive also the manualised Cognitive Behaviour Therapy treatment for Panic Disorder, delivered in the outpatient psychotherapy centre of the Department of Clinical Psychology and Psychotherapy, Ruhr-Universität Bochum.
- Anxious Control Group: CBT (Other): All participants in the Anxious Control Group will receive a manualised Cognitive Behaviour Therapy (CBT) treatment for their diagnosed anxiety disorder, delivered in the outpatient psychotherapy centre of the Department of Clinical Psychology and Psychotherapy, Ruhr-Universität Bochum.
  Interventions: Behavioral: Cognitive Behaviour Therapy

INTERVENTIONS:
Behavioral: Cognitive Behaviour Therapy — Cognitive Behaviour Therapy (CBT) for diagnosed anxiety disorder (i.e. CBT for Panic Disorder in the Panic Disorder group, or other diagnosed anxiety disorders in the Anxious Control group.
  Arms: Anxious Control Group: CBT; Panic Disorder: CBT

SUMMARY:
The aim of the study is to examine panic-related associations and interpretations in the context of Panic Disorder and its treatment. While theoretical accounts of Panic Disorder suggest a central role of such associations and interpretations in the onset and maintenance of the disorder, research to date in fact leaves many questions about the nature of these dysfunctional cognitions and their potential role unanswered. Patients with Panic Disorder and a control group of patients with other anxiety disorders will complete measures of panic-relevant associations and interpretation bias. The patients with Panic Disorder will be randomized to receive either Cognitive Behaviour Therapy (CBT) or a waiting list condition (to be followed by CBT after completion of the study procedures). The anxious control group will also receive CBT. Panic-relevant associations and interpretations will be measured twice, i.e., pre and post CBT/waitlist. Furthermore, relevant symptom measures and physiological and biological markers will be assessed and responses to a hyperventilation challenge. The study aims to further advance our understanding of cognitions in the etiology and maintenance of Panic Disorder, and inform future treatment optimisation.

DETAILED DESCRIPTION:
The main purpose of the present study is to look at relationships and changes over time but not to compare treatment outcomes (i.e. it is not an efficacy trial). The associations and interpretation measures are listed as primary outcomes because these are the measures of main interest.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65
* Primary DSM-5 Anxiety Disorder (Panic Disorder for Panic Disorder groups, other anxiety disorder for anxious control group)
* Provided written informed consent
* Patient is in principle able to take part in the therapy
* Sufficient knowledge of German language
* Outpatient (no parallel hospital stay)
* Medical certificate: medical safety, so that hyperventilation is possible

Exclusion Criteria:

* Any reason that jeopardises the performance of the therapy
* Acute suicidality
* Primary affective disorder (e.g. Bipolar I, Major Depression)
* Psychotic disorder
* Parallel psychiatric or psychotherapeutic treatment (acute treatment)
* Current substance dependence (apart from Nicotine dependence)
* Serious medical disorders/ findings
* Other primary treatment diagnosis
* Intellectual impairment (estimated during screening)
* ADHD (estimated during screening)
* Personality disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Priming Task | Change from pre-treatment/waitinglist - post-treatment/waitinglist (post is approx. 3 months after the pre-treatment/waitinglist assessment)
  The Priming Paradigm measures panic related associations. During this task, participants will be instructed to sort target words as words versus non-words (lexical decision task). Before a target appears, however, a prime will be presented. Participants will be instructed to look at the prime but to not react to it. Following the design of Hermans et al. (2010), we will use the following prime-target combinations: panic-panic, panic-neutral, neutral-neutral, neutral-panic. There will also be prime-target combinations with non-words as targets.
Single Target Association Test | Change from pre-treatment/waitinglist - post-treatment/waitinglist (post is approx. 3 months after the pre-treatment/waitinglist assessment)
  The Single Target Implicit Association Test (STIAT) measures the associative strength between a target concept and two attribute dimensions. Participants are asked to sort stimuli into three categories by means of two response keys: one category represents a target concept, and two categories represent two poles of an attribute dimension. The target category is paired with both attributes. The present STIAT is designed as follows: targets: bodily changes, attributes: alarming vs. meaningless, and it takes over the structure as suggested by Wigboldus et al. (2006): (a) attribute discrimination, (b) target categorization practice, (c) first combined block, (d) reversed target categorization practice, and (e) reversed combined block.
Scrambled Sentences Test | Change from pre-treatment/waitinglist - post-treatment/waitinglist (post is approx. 3 months after the pre-treatment/waitinglist assessment)
  The Scrambled Sentence Task (SST, Wenzlaff & Bates, 1998) measures panic-related interpretation biases. It consists of six-word strings participants are asked to unscramble to form a five-word sentence, leaving out one word. The present SST can be completed such that the resulting five-word sentences produce either a panic-related or neutral interpretation. During the SST, there is a cognitive load, i.e., participants have to memorize a 6 digit number.
Interpretation Bias Questionnaire | Change from pre-treatment/waitinglist - post-treatment/waitinglist (post is approx. 3 months after the pre-treatment/waitinglist assessment)
  The Interpretation Bias Questionnaire (IBQ) measures panic-related interpretation biases. It consists of 18 brief scenarios used in earlier studies (Ebert, 1993, Foa & McNally, 1987). Nine items describe panic-related situations, and the other nine describe negative, threat-related situations. Following each scenario, three explanations are presented (for panic-related scenarios: one panic-related explanation and two panic-unrelated explanations, for negative, threat-related situations: one very negative, threat-related interpretation and two harmless explanations). Participants have to indicate how likely each explanation for the corresponding scenario is, using rating scale from 0 (not likely) to 100 (very likely).

SECONDARY OUTCOMES:
Anxiety Sensitivity Index (ASI) | Pre-treatment/waitinglist - post-treatment/waitinglist (post is approx. 3 months after the pre-treatment/waitinglist assessment)
  The ASI (Ehlers, 1986; Reiss, Peterson, & McNally, 1986) is a 16-item self-report questionnaire measuring fear and concerns regarding anxiety-related symptoms such as "It scares me when my heart beats rapidly". Items are rated on a five-point Likert scale (0 = "Very little" to 4 = "Very much").
Depression Anxiety Stress Scale (DASS) | Pre-treatment/waitinglist - post-treatment/waitinglist (post is approx. 3 months after the pre-treatment/waitinglist assessment)
  The DASS-21 (Lovibond & Lovibond, 1995; Nilges & Essau, 2015) questionnaire comprises three 7-item subscales assessing levels of depression, anxiety, and stress.
Agoraphobic Cognitions Questionnaire (ACQ) | Pre-treatment/waitinglist - post-treatment/waitinglist (post is approx. 3 months after the pre-treatment/waitinglist assessment)
  The ACQ (Chambless, Caputo, Bright, & Gallagher, 1984; Ehlers, Margraf, & Chambless, 1993) measures maladaptive thoughts about the potential for disastrous consequences arising from anxiety or panic. It includes 14 items which can be scored as a total scale, or according to its two subscales, "loss of control" and "physical concerns".
Body Sensations Questionnaire (BSQ) | Pre-treatment/waitinglist - post-treatment/waitinglist (post is approx. 3 months after the pre-treatment/waitinglist assessment)
  The BSQ (Chambless, Caputo, Bright, & Gallagher, 1984; Ehlers, Margraf, & Chambless, 1993) includes 17 items that reflect specific bodily sensations (e.g., heart palpations, dizziness). Participants are asked to indicate the degree to which they experience anxiety related to these sensations by means of a five-point Likert scale (1 = "Not at all" to 5 = "Extremely").
Panic Disorder Severity Scale (PDSS) | Pre-treatment/waitinglist - post-treatment/waitinglist (post is approx. 3 months after the pre-treatment/waitinglist assessment)
  The PDSS (Shear et al., 1997) is a 7-item scale and provides a composite severity score of frequency, distress, and impairment associated with panic attacks.
Mobility Inventory (MI) | Pre-treatment/waitinglist - post-treatment/waitinglist (post is approx. 3 months after the pre-treatment/waitinglist assessment)
  The MI (Chambless, Caputo, Jasin, Gracely, & Williams, 1985, Ehlers, Margraf, & Chambless, 1993) consists of 26 items and measures agoraphobic avoidance using a five-point Likert scale (1 = "Never avoid" to 5 = "Always avoid"). Each item has to be answered twice, once for when being accompanied and once for when being alone.
Subjective ratings DSM panic symptoms | Pre-treatment/waitinglist - post-treatment/waitinglist (post is approx. 3 months after the pre-treatment/waitinglist assessment)
  A symptom checklist will assess the presence of panic-relevant symptomatology in line with the DSM-5 criteria for panic disorder, e.g., occurrence and frequency of panic attacks, experienced distress during panic attack, fear of going crazy, dizziness etc. (for a similar procedure, see Wilhelm, Gerlach, & Roth, 2001). It also assess participants' level of generally anxiety and whether or not participants experienced a panic attack. This will be completed repeatedly within each testing session.
Responses Hyperventilation Task | Pre-treatment/waitinglist - post-treatment/waitinglist (post is approx. 3 months after the pre-treatment/waitinglist assessment)
  An adapted version of the procedure described by Kossowsky, Wilhelm, and Schneider (2013) and Wilhelm et al. (2001) will be used in the present study. During the hyperventilation, participants will breathe through their nose and their breathing will be monitored by a capnograph. There will be 3 phases.
  Phase 1: Participants will undergo a 'paced breathing' procedure. That is, they will be asked to keep a breathing speed of 18 cycles/minute (breaths per minute, bpm). Breathing speed will be paced by computerized audio instructions. At the end of phase 1, the end-tidal CO2 level should be 25mmHg (for recommendations for the end-tidal level, see Meuret et al., 2005).
  Phase 2: The goal of this phase is to maintain the 25mmHg CO2 level while participants keep on breathing with a 18 bpm paced breathing pattern.
  Phase 3: This is a 3 minute recovery phase. During this phase, participants are supposed to breath normally again.
Heart rate variability | Pre-treatment/waitinglist - post-treatment/waitinglist (post is approx. 3 months after the pre-treatment/waitinglist assessment)t
  An Electrocardiogram (ECG) will assess heart rate variability (HRV) during each testing session
Muscle activity | Pre-treatment/waitinglist - post-treatment/waitinglist (post is approx. 3 months after the pre-treatment/waitinglist assessment)
  An Electromyography (EMG) will assess facial muscle activity during each testing session.
Respiration | Pre-treatment/waitinglist - post-treatment/waitinglist (post is approx. 3 months after the pre-treatment/waitinglist assessment)
  Following recommendations of Ritz and Dahme (2006), the HRV assessment will be combined with a respiratory assessment. Respiration will be assessed by means of two plethysmography belts (thorax and abdomen) during each testing session.
Galvanic skin response | Pre-treatment/waitinglist - post-treatment/waitinglist (post is approx. 3 months after the pre-treatment/waitinglist assessment)
  Electrodermal activity (EDA), i.e., variations in the electrical characteristics of the skin, will be assessed during each testing session.
Cortisol | Pre-treatment/waitinglist - post-treatment/waitinglist (post is approx. 3 months after the pre-treatment/waitinglist assessment)
  Saliva samples will be collected at the start, during, and at the end of each testing session to analyze changes in cortisol levels, which serve as indices of arousal and stress.
Alpha amylase | Pre-treatment/waitinglist - post-treatment/waitinglist (post is approx. 3 months after the pre-treatment/waitinglist assessment)
  Saliva samples will be collected at the start, during, and at the end of each testing session to analyze changes in alpha amylase, which serve as indices of arousal and stress.

CONTACTS AND LOCATIONS:
Overall Officials: Marcella L Woud, PhD, Principal Investigator — Ruhr University of Bochum
Locations (1):
- Psychotherapy Centre, Department of Clinical Psychology and Psychotherapy, Ruhr-Universität Bochum, Bochum, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
It is planned to make individual participant data available on publication of the associated study results, via a publically-available data repository such as Open Science Framework. Data made available will be the research data reported in the publication, with the exception of any data that could compromise participant anonymity.